CLINICAL TRIAL: NCT04137354
Title: Effects of Intermittent Iron and Vitamin A Supplementation on Nutritional Status and Development of Schoolchildren in Arba Minch Zuria District, Ethiopia.
Brief Title: Iron and Vitamin A in School Children
Acronym: IronVitA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Flemish Interuniversity Council (VLIR) (Network); Arba Minch University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EC/2019/1289
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Anemia, Iron Deficiency; Vitamin A Deficiency; Cognitive Development; Helminthic Infection
Keywords: Intermittent Iron supplementation; Vitamin A; Cognitive Development; Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Vitamin A Deficiency; Trematode Infections; Anemia

STUDY DESIGN:
Intervention Model Description: In randomized placebo-control trial eligible primary school children in the Arba Minch HDSS will be randomly assigned to four groups of treatment in a factorial 2x2 design:
  1. A control placebo receiving placebo vitamin A at baseline and after 5 months, and placebo iron supplement weekly;
  2. A high dose vitamin A at baseline and after 5 months and weekly placebo iron supplement;
  3. Weekly iron supplementation for 10 months and placebo vitamin A at baseline and after 5 months;
  4. Combined weekly iron supplementation and high dose vitamin A at baseline and after 5 months.
  At the end of the study, and if the results are positive, children who receive the placebo iron supplement will receive weekly iron supplementation (42mg of elemental iron once a week) for 10 months. Children in all the treatment groups remain eligible to benefit from the standard health care and nutrition programs provided at school, such as deworming at the beginning of the school year
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Iron supplements and their placebo: Both iron and placebo supplements will be produced by Metagenics (Belgium) for the context of this study. Placebo tablets will have the same taste, and shape of the iron tablets, the colour is slightly different because of the characteristics of the products but the blinding is ensured. The blister/ the tablets will be packed and only coded.
  Vitamin A and its placebo: Vitamin A capsule is oral liquid, red, oil-based preparation of retinyl palmitate that contains the equivalent of 100,000 IU (110μmol) of vitamin A and stabilized with 20IU of vitamin E. The placebo supplement will have the same oil composition except that it will not contain vitamin A equivalent. Placebo oil and vitamin A preparation will be transferred to two colored (red and orange) Eppendorf® Safe-Lock microcentrifuge tubes volume 0.6 mL by a researcher who is not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Iron&Vitamin A Placebo (Placebo Comparator): Children randomly assigned to the placebo iron & vitamin A control group will receive weekly three placebo tablets that are identical to the iron tablets (blinded) for the whole duration of the study (9 months of the school year). They will also receive placebo vitamin A at baseline and at mid-line (after 4.5 months).
  Interventions: Other: Intermittent placebo iron supplement; Other: Placebo Vitamin A
- Vitamin A & Placebo Iron Supplements (Experimental): Children is this group will receive weekly three placebo tablets that are identical to the iron tablets (blinded) for the whole duration of the study (9 months of the school year). They will also receive a high dose vitamin A capsule (200,000IU) at baseline and after 4.5 months (at mid-line)
  Interventions: Other: Intermittent placebo iron supplement; Other: High-dose Vitamin A supplement
- Intermittent Iron Supplements & Placebo Vitamin A (Experimental): Children is this group will receive weekly three tablets of iron (42mg of elemental iron once a week) for 9 months (equivalent to a one school year).
  They will also receive placebo vitamin A at baseline and at mid-line (after 4.5 months).
  Interventions: Other: Intermittent iron supplement; Other: Placebo Vitamin A
- Intermittent Iron Supplements & High dose Vitamin A (Experimental): Combined weekly iron supplementation (42mg of elemental iron once a week) for 9 months and high dose vitamin A (200,000IU) at baseline and after 4.5 months (mid-line).
  Interventions: Other: Intermittent iron supplement; Other: High-dose Vitamin A supplement

INTERVENTIONS:
Other: Intermittent placebo iron supplement — Placebo iron supplements are also three tablets containing the same ingredients as for iron tablets and will be given to the children on a weekly basis for the whole duration of the intervention (i.e. the school year of 9 months)
  Other Names: Control iron
  Arms: Control Iron&Vitamin A Placebo; Vitamin A & Placebo Iron Supplements
Other: Intermittent iron supplement — Three iron tablets containing 42 mg of elemental iron will be provided to the children on a weekly basis for the whole duration of the intervention (i.e. the school year of 9 months)
  Other Names: Experimental iron
  Arms: Intermittent Iron Supplements & High dose Vitamin A; Intermittent Iron Supplements & Placebo Vitamin A
Other: Placebo Vitamin A — Children will receive in a colorful Eppendorf tube 400 micro-liter of corn oil stabilized with vitamin A twice during the intervention period of 9 months, at baseline (after enrollment) and at mid-line (4.5 months).
  Other Names: Control Vitamin A
  Arms: Control Iron&Vitamin A Placebo; Intermittent Iron Supplements & Placebo Vitamin A
Other: High-dose Vitamin A supplement — Children will receive in a colorful Eppendorf tube 400 micro-liter of oil-based preparation of retinyl palmitate that contains the equivalent of 100,000 IU (110μmol) of vitamin A and stabilized with 20IU of vitamin E twice during the intervention period of 9 months, at baseline (after enrollment) and at mid-line (4.5 months).
  Other Names: Experimental Vitamin A
  Arms: Intermittent Iron Supplements & High dose Vitamin A; Vitamin A & Placebo Iron Supplements

SUMMARY:
The WHO recommended intermittent iron supplementation as a strategy for prevention of anemia and iron deficiency among school age children. Several aspects of cognitive development, co-supplementation with other micronutrients, severe adverse events especially in the context of malaria were missing.

The investigators will evaluate the effectiveness of intermittent iron and vitamin A supplementation on cognitive development and anemia and iron status of Rural Ethiopian school children.

DETAILED DESCRIPTION:
Iron deficiency is the commonest micronutrient deficiency worldwide and the major cause of specific anemia - iron deficiency anemia. Iron is an essential mineral with lots of functions in the human body; its deficiency is associated with cognitive impairment, emotional alteration, and altered homeostasis in myelination and neurotransmission. Vitamin A deficiency can lead to anemia, weakened resistance to infection, blindness, and death. Animal model studies showed that vitamin A could affect cognition. Cognitive skills, influenced by cognitive development of the individual, are related with academic performance of the student and long-term success. One target of the Sustainable Development Goals (SDG 4) is to ensure inclusive and equitable quality education and promote lifelong learning opportunities for all. Poor health and undernutrition of children in Low- and Middle-Income Countries (LMIC) are the major limitations to reach their potential school performance and learning skills. The evidence on the role of intermittent iron supplementation in preventing anemia is strong but several aspects of cognitive development, co-supplementation with other micronutrients such as vitamin A are missing.

The aim of this study is to evaluate the effectiveness of intermittent iron and high-dose vitamin A supplementation integrated within school nutritional plan on anemia, iron status and cognitive development of school children (7 - 10 year old) who live in areas with high rates of food insecurity in Ethiopia.

Method: The study will be carried out at primary schools in Arba Minch Zuria District, Ethiopia in children aged from 7 to 10 years. Eligible children (a total of 504 children) will be randomly assigned to one of the four groups: 1) Control placebo receiving placebo vitamin A and placebo iron supplement; 2) Vitamin A group will receive a high dose vitamin A capsule (200,000 IU) and placebo iron supplement.;3) Iron group will receive weekly iron supplementation (42 mg of elemental iron) and placebo vitamin A; and 4)Iron-vitamin A group will receive a combined weekly iron supplementation and high dose vitamin A.

Iron supplements (42mg of elemental iron)/placebo will be given to school chidlren weekly for 10 months and 200,000 IU of vitamin A/placebo will be given at baseline and after 5 months.

ELIGIBILITY:
Inclusion Criteria:

* One or both their parents signed informed consent form;
* Their parents planned to stay during the period of the study (for the full academic year) in the kebele; and
* They accept of the intervention package including blood draw and home visits. School children with severe anemia (Hb concentration <80 g/L) will be treated by conventional protocol for three months at nearby health centres. After reassessing their haemoglobin concentrations, they can be assigned to their intervention groups if they become eligible as described above.

Exclusion Criteria:

* Chronically ill children like diagnosed diabetic and asthma
* Severely under nourished children (defined as body mass index z-score <-3 standard deviations of the median WHO reference population)
* Those who are treated for tuberculosis or suspected to have tuberculosis
* Children with diagnosed haemoglobinopathy (sickle cell and thalassemias)
* Children with night blindness

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 504 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Memory span | Memory span of the children will be assessed at 9 months
  Digit span (forward and backward) is a standardized test that assess the working memory of the children, one indicator of cognitive development
Spatial exploration and awareness | Spatial exploration and awareness of the children will be assessed at 9 months
  Vision search using cancellation task of the children, the second indicator of cognitive development
Reasoning ability | The reasoning ability of the children will be assessed at 9 months
  Raven's colored progressive matrices, the third indicator of cognitive development
Anemia | Hemoglobin concentrations of children will be assessed at 9 months
  Hemoglobin concentrations (g/dL)
Plasma ferritin | Plasma ferritin is assessed in all children at 9 months
  Iron status as indicated plasma ferritin (micro_g/L) is a test to evaluate iron stores
Soluble transferrin receptor | Soluble transferrin receptor is assessed in all children at 9 months
  Soluble transferrin receptor (mg/L) is an indicator for iron deficiency especially in high inflammation settings

SECONDARY OUTCOMES:
Serum concentrations in Vitamin A (retinol) | Retinol concentrations will be assessed in all children at 9 months
  Retinol concentrations in serum is an indicator of vitamin A status of children
Serum concentrations in vitamin B12 | Vitamin B12 concentrations will be assessed in all children at 9 months
  Serum concentrations in vitamin B12
Prevalence of soil-transmitted helminths | The prevalence of soil-transmitted helminths will be assessed at 4.5 months and at 9 months
  The presence of worm parasites and egg density in the stools. Three common parasites and their eggs will be investigated, i.e. Ascaris lumbricoides (round worm), Trichuris trichiura (whipworm) and Ancyclostoma duodenale or Necater americanus (hookworms).
Prevalence of Schistosome infection | Prevalence of Schistosome infection will be assessed at 4.5 months and at 9 months
  The prevalence of Schistosoma mansoni infection
Adherence to the iron/placebo supplements | Weekly for the whole period of the intervention of 9 months.
  Adherence to the tablets of Iron/Placebo will be assessed through teacher's reports. Teachers are the ones who are providing the supplements in a weekly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent
Locations (1):
- Arba Minch University, Arba Minch, Ethiopia

IPD SHARING:
Plan to Share IPD: No
All the data that can affect the main or the secondary outcomes will be used in the analyses and shared as necessary.
  Data on helminthic infection will use characteristics of the attended schools, villages and of the child (date of birth).

REFERENCES:
- [Background] Guideline: Intermittent Iron Supplementation in Preschool and School-Age Children. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK179850/ PMID 24479203
- [Background] De-Regil LM, Jefferds ME, Sylvetsky AC, Dowswell T. Intermittent iron supplementation for improving nutrition and development in children under 12 years of age. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD009085. doi: 10.1002/14651858.CD009085.pub2. PMID 22161444
- [Background] Friis H, Mwaniki D, Omondi B, Muniu E, Magnussen P, Geissler W, Thiong'o F, Michaelsen KF. Serum retinol concentrations and Schistosoma mansoni, intestinal helminths, and malarial parasitemia: a cross-sectional study in Kenyan preschool and primary school children. Am J Clin Nutr. 1997 Sep;66(3):665-71. doi: 10.1093/ajcn/66.3.665. PMID 9280190
- [Background] Zimmermann MB, Biebinger R, Rohner F, Dib A, Zeder C, Hurrell RF, Chaouki N. Vitamin A supplementation in children with poor vitamin A and iron status increases erythropoietin and hemoglobin concentrations without changing total body iron. Am J Clin Nutr. 2006 Sep;84(3):580-6. doi: 10.1093/ajcn/84.3.580. PMID 16960172
- [Background] Mwaniki D, Omondi B, Muniu E, Thiong'o F, Ouma J, Magnussen P, Geissler PW, Michaelsen KF, Friis H. Effects on serum retinol of multi-micronutrient supplementation and multi-helminth chemotherapy: a randomised, controlled trial in Kenyan school children. Eur J Clin Nutr. 2002 Jul;56(7):666-73. doi: 10.1038/sj.ejcn.1601376. PMID 12080408
- [Derived] Gutema BT, Tariku EZ, Melketsedik ZA, Levecke B, De Henauw S, Abubakar A, Abbeddou S. Assessing the influence of COVID-19 lockdown measures on cognition and behavior in school age children in Arba Minch Health and Demographic Surveillance site, Southern Ethiopia: A cross-sectional study. PLOS Glob Public Health. 2024 Mar 21;4(3):e0002978. doi: 10.1371/journal.pgph.0002978. eCollection 2024. PMID 38512931
- [Derived] Gutema BT, Levecke B, Sorrie MB, Megersa ND, Zewdie TH, Yesera GE, De Henauw S, Abubakar A, Abbeddou S. Effectiveness of intermittent iron and high-dose vitamin A supplementation on cognitive development of school children in southern Ethiopia: a randomized placebo-controlled trial. Am J Clin Nutr. 2024 Feb;119(2):470-484. doi: 10.1016/j.ajcnut.2023.11.005. Epub 2023 Nov 11. PMID 37952928